CLINICAL TRIAL: NCT06305507
Title: Effects of Differents Laser Applications on Plantar Fasciitis
Brief Title: Differents Laser Applications on Plantar Fasciitis
Acronym: FASLaser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Profesor Titular Doctor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30923-N
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Fasciitis, Plantar
Keywords: Fascitis Plantar; Focused laser therapy; Randomized Clinical trial; Doubled blinded; Longitudinal; Pain reduction; Therapeutic; Session duration; Comparision group
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Magnetic Field Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Pilot Study with Two Parallel Groups. Participants were randomly assigned to one of two experimental groups (High-Intensity Laser Therapy in Static Mode or High-Intensity Laser Therapy in Scanning Mode) to receive 12 treatment sessions over a 40-day period. This is a single-blind design, where participants were blinded to the type of laser application received.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT Static mode (Other): Hilt Scanning mode
  Interventions: Other: Static therapy
- Shower laser application (Active Comparator): laser application in shower or sweep mode
  Interventions: Other: Static Mode

INTERVENTIONS:
Other: Static therapy — The intervention involves the precise and focused application of HILT on specific areas related to plantar fasciitis. The static mode technique is characterized by directing the laser directly to the painful point, seeking optimal stimulation in the affected region.The Scanning Mode technique is characterized by applying the HILT through a continuous, sweeping movement of the handpiece over the target area
  Arms: HILT Static mode
Other: Static Mode — The Scanning Mode technique is characterized by applying the HILT through a continuous, sweeping movement of the handpiece over the target area (the plantar fascia and adjacent tender regions).
  This application ensures a more uniform energy distribution across a larger tissue area, potentially addressing inflammation and pain in a broader region than the static mode. The total dose is distributed over the area treated with a continuous motion.
  Other Names: Sweeping laser therapy
  Arms: Shower laser application

SUMMARY:
The objective of this randomized controlled clinical trial (RCT) with a double-blind technique and longitudinal chronology, is to evaluate and compare the effectiveness of High intensity laser therapy (HILT) in static mode versus scanning mode in the reduction of pain associated with plantar fasciitis.

The main questions it seeks to answer are:

* What is the comparative effectiveness between low-level laser therapy in local spot mode and sweep mode in reducing pain in patients with plantar fasciitis?
* What are the optimal therapeutic parameters (session duration, frequency and power) for LLLT in both modes, maximizing pain reduction in patients with plantar fasciitis?

Participants in this study will perform the following tasks:

* Undergo HILT sessions or scanning mode.
* Comply with the instructions on the duration and frequency of the sessions.
* Record the pain levels experienced before and after each session.

The investigators will compare the group this differents laser to evaluate whether there are significant differences in pain reduction effects.

DETAILED DESCRIPTION:
This randomized controlled clinical trial, titled 'Effect of Different Laser Applications on Plantar Fasciitis', aims to specifically address the effectiveness of static mode versus scanning mode (HILT) in the treatment of pain associated with plantar fasciitis. Using a rigorous methodology that includes double-blind masking and a longitudinal chronology, the study focuses on comparing two modes of laser application.

The main objective is to evaluate and compare the pain reduction between these two modes of application of LLLT. To achieve this, key questions are asked, such as the relative effectiveness of each mode and the identification of optimal therapeutic parameters, including session duration, frequency and power, that maximize benefits in patients with plantar fasciitis.

Participants in this study will undergo low-level laser therapy sessions, following the protocols established for each mode of application. Additionally, they will be asked to record their pain levels before and after each session, providing valuable information about the effectiveness of the therapy.

In the case of a comparison group, a detailed evaluation will be carried out comparing the results obtained between the group treated with static in local spot mode and the group treated in scanning mode. This approach will allow researchers to determine if there are significant differences in the pain reduction effects between the two modes of laser application.

With a solid experimental design and specific objectives, this study seeks to contribute significantly to the understanding of laser applications in the treatment of plantar fasciitis, providing valuable information for the optimization of therapy and thus improving the quality of life of patients. . affected.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of Plantar Fasciitis (at least 8 weeks), adults,

Exclusion Criteria:

* Additional Serious Medical Conditions, Not receiving treatment at the time of the study for plantar fasciitis, neither, serious disease, a score of >3 on the DN4 questionnaire neuropathic pain, neither Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Visual pain analogic scale | 1,2 and 4 months
  Visual pain scale from 0 minimum (best) to 10 maximum (worse)

SECONDARY OUTCOMES:
Ultrasound image of thickness | 1,2 and 4 months
  fascia thickness measured by ultrasound from minumum of 3 (Best) to maximum of 6 mm (Worse)

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Castro Mendez, PhD, Principal Investigator — University of Seville
Locations (2):
- Spain (2):
  - Área Clínica de Podología, Seville, Andalusia
  - Fasciitis, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guimaraes JS, Arcanjo FL, Leporace G, Metsavaht LF, Sena C, Moreno MVMG, Marcal Vieira TE, Gomes Neto M. Effect of low-level laser therapy on pain and disability in patients with plantar fasciitis: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2022 Feb;57:102478. doi: 10.1016/j.msksp.2021.102478. Epub 2021 Nov 16. PMID 34847470
- [Result] Takla MKN, Rezk SSR. Clinical effectiveness of multi-wavelength photobiomodulation therapy as an adjunct to extracorporeal shock wave therapy in the management of plantar fasciitis: a randomized controlled trial. Lasers Med Sci. 2019 Apr;34(3):583-593. doi: 10.1007/s10103-018-2632-4. Epub 2018 Sep 7. PMID 30194553
- [Result] Kiritsi O, Tsitas K, Malliaropoulos N, Mikroulis G. Ultrasonographic evaluation of plantar fasciitis after low-level laser therapy: results of a double-blind, randomized, placebo-controlled trial. Lasers Med Sci. 2010 Mar;25(2):275-81. doi: 10.1007/s10103-009-0737-5. PMID 19841862